CLINICAL TRIAL: NCT04189224
Title: Clinical Evaluation of a Reusable Multifocal Optical Design in a Presbyopic Population Phase II
Brief Title: Evaluation of a Reusable Silicone Hydrogel Multifocal Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-6372
Record Dates: First submitted 2019-12-04; First posted 2019-12-06 (Actual); Results first posted 2021-04-02 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Test/Control (Experimental): Hyperopic subjects that are habitual soft contact lens wearers and have presbyopia will be randomized to sequence, Test/Control.
  Interventions: Device: JJV Investigational Multifocal Contact Lens; Device: 1-Day Acuvue® Moist Brand Multifocal Contact Lens
- Control/Test (Experimental): Hyperopic subjects that are habitual soft contact lens wearers and have presbyopia will be randomized to sequence, Control/Test.
  Interventions: Device: JJV Investigational Multifocal Contact Lens; Device: 1-Day Acuvue® Moist Brand Multifocal Contact Lens

INTERVENTIONS:
Device: JJV Investigational Multifocal Contact Lens — TEST
Device: 1-Day Acuvue® Moist Brand Multifocal Contact Lens — CONTROL

SUMMARY:
This study is a randomized, single-masked, crossover clinical trial. There are two study lenses. Each lens will be dispensed for 3 ± 1 days and then an optimization visit will occur. The final lens pair will be dispensed for 12 ± 2 days and the follow-up on the final lens pair will occur. The second study lenses will then be fit and the above sequence repeated.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following criteria to be enrolled in the study:

  1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
  2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
  3. The subject must be at least 40 years of age and not greater than 70 years of age at the time of consent.
  4. Subjects must own a wearable pair of spectacles if required for their distance vision.
  5. The subject must be an adapted soft contact lens wearer in both eyes (i.e. worn lenses a minimum of 2 days per week for at least 8 hours per wear day, for 1 month or more duration).
  6. The subject must either already be wearing a presbyopic contact lens correction (e.g., reading spectacles over contact lenses, multifocal or monovision contact lenses, etc.) or if not respond positively to at least one symptom on the "Presbyopic Symptoms Questionnaire" (Appendix E).
  7. The subject's distance spherical equivalent refraction must be in the range of +1.25 D to +3.75 D in each eye.
  8. The subject's refractive cylinder must be ≤0.75 D in each eye.
  9. The subject's ADD power must be in the range of +0.75 D to +2.50 D.
  10. The subject must have distance best corrected visual acuity of 20/20-3 or better in each eye.

      Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Currently pregnant or lactating.
  2. Any active or ongoing ocular or systemic allergies that may interfere with contact lens wear.
  3. Any active or ongoing systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear. This may include, but not be limited to, diabetes, hyperthyroidism, Sjögren's syndrome, xerophthalmia, acne rosacea, Stevens- Johnson syndrome, and immunosuppressive diseases or any infectious diseases (e.g. hepatitis, tuberculosis).
  4. Any previous, or planned, ocular or intraocular surgery (e.g. radial keratotomy, PRK, LASIK, lid procedures, cataract surgery, retinal surgery, etc.).
  5. A history of amblyopia, strabismus or binocular vision abnormality.
  6. Use of any of the following medications within 1 week prior to enrollment: oral retinoid isotretinoin (e.g. Accutane), oral tetracyclines, oral phenothiazines, oral/topical/inhaled anticholinergics, systemic/topical corticosteroids.
  7. Use of any ocular medication, with the exception of rewetting drops.
  8. History of herpetic keratitis.
  9. History of irregular cornea.
  10. History of pathological dry eye.
  11. Participation in any contact lens or lens care product clinical trial within 30 days prior to study enrollment.
  12. Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
  13. Any known hypersensitivity or allergic reaction to Optifree®Replenish® multipurpose care solution, sodium fluorescein or non-preserved rewetting drop solutions.
  14. Clinically significant (Grade 2 or greater) corneal edema, corneal vascularization, corneal staining, tarsal abnormalities or bulbar injection, or any other corneal or ocular abnormalities which would contraindicate contact lens wear.
  15. Entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions.
  16. Any current ocular infection or inflammation.
  17. Any current ocular abnormality that may interfere with contact lens wear.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Maitland Vision Center, Maitland, Florida
  - Advanced Eyecare, Raytown, Missouri
  - ProCare Vision Centers, Granville, Ohio
  - Frazier Vision Inc., Jacksonville, Texas

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 46 subjects were enrolled in this study. Of those enrolled, 44 (95.7%) subjects randomized and dispensed at least 1 study lens while, 2 (4.3%) subjects failed to meet all eligibility criteria. Of those dispensed, 43 (93.5%) subjects completed the study while, 1 (2.2%) subject was discontinued from the study.
Groups:
- Test/Control: Subjects randomized to this sequence received the Test lens during the first period and then received the Control lens during the second period.
- Control/Test: Subjects randomized to this sequence received the Control lens during the first period and then received the Test lens during the second period.
Period: Period 1
Arm/Group | Test/Control | Control/Test
Started | 23 | 21
Completed | 23 | 21
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Test/Control | Control/Test
Started | 23 | 21
Completed | 23 | 20
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: All subjects dispensed a study lens.
Groups:
- All Participants: Subjects that wore either Test or Control lens in either first or second period of the study.
Arm/Group | All Participants
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (6.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 43
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Binocular Contact Lens-Corrected Visual Performance Under Standard High Contrast Bright
Description: The contact lens-corrected visual performance on logMAR scale was evaluated binocularly under high luminance high contrast, dim luminance high contrast and high luminance low contrast conditions at 4 meters (distance), 64 cm (intermediate) and 40 cm (near) using ETDRS/reduced Guillon-Poling charts. A value of 0.0 logMAR equates to 20/20 vision on a Snellen Scale. Lower values indicate better visual performance. The average visual performance was reported for each lens type and distance.
Time Frame: 2-Week Follow-up
Population: Analysis population consisted of all subjects who had successfully completed the study and did not substantially deviate from the protocol.
Measure: Mean (Standard Deviation); unit: logMAR
Groups:
- Test (Senofilcon A): Subjects that wore the Test lens in either the first or second period of the study.
- Control (Etafilcon A): Subjects that wore the Control lens in either the first or second period of the study.
Arm/Group | Test (Senofilcon A) | Control (Etafilcon A)
Number analyzed (Participants) | 40 | 40
logMAR
  Standard High Contrast Bright: Distance | -0.12 (0.073) | -0.12 (0.067)
  Standard High Contrast Bright: Intermediate | -0.06 (0.070) | -0.06 (0.072)
  Standard High Contrast Bright: Near | 0.07 (0.097) | 0.08 (0.106)

2. Secondary Outcome: Overall Vision Scores
Description: Overall vision scores were assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, aged 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120.
Time Frame: 2-Week Follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: CLUE points
Arm/Group | Test (Senofilcon A) | Control (Etafilcon A)
Number analyzed (Participants) | 40 | 40
CLUE points | 52.24 (22.035) | 50.24 (23.282)

3. Secondary Outcome: Overall Comfort Scores
Description: Overall comfort scores were assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, aged 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120.
Time Frame: 2-Week Follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: CLUE points
Arm/Group | Test (Senofilcon A) | Control (Etafilcon A)
Number analyzed (Participants) | 40 | 40
CLUE points | 64.51 (26.630) | 62.71 (24.006)

4. Secondary Outcome: Number of Grade 3 or Higher Slit Lamp Findings
Description: Slit Lamp Findings (SLF) were assessed using a biomicroscope and was graded using the FDA grading scale (Grade: 0, 1,2, 3 and 4) with grade 0 represents the absence of findings and 1 to 4 representing successively worse findings (i.e. Grade 1 = trace, Grade 2 = Mild, Grade 3 = moderate and Grade 4 = severe). Slit Lamp Findings were assessed at the 2-Week Follow-up. SLF is a binary response where Y=1 for at least one Grade 3 or 4 slit lamp finding. The number of eyes with SLF with grade 3 or higher by lens was reported.
Time Frame: 2-Week Follow-up
Population: Analysis population consisted of all subjects who were dispensed at least 1 study lens.
Measure: Number; unit: number of eyes
Units Other Than Participants: number of eyes
Arm/Group | Test (Senofilcon A) | Control (Etafilcon A)
Number analyzed (Participants) | 44 | 44
Number analyzed (number of eyes) | 88 | 88
number of eyes | 0 | 0

5. Secondary Outcome: Proportion of Subjects That Reported Ocular Symptoms
Description: Subject reported ocular symptoms were assessed using a questionnaire at the 2-week follow-up. Subjects were asked if they experienced any of the following symptoms: Burning/Stinging, Itchiness/Scratchiness, Dryness, Lens Awareness, Grittiness/Foreign Body Sensation, Redness, Irritation/Discomfort, Cloudy/Blurry/Hazy, Variable Vision and Other; using the scale of: None, Mild, Moderate and Severe. The proportion of subjects that reported symptoms (Mild, Moderate and Severe) was reported for each lens type.
Time Frame: 2-Week Follow-up
Population: Analysis population consisted of all subjects who were dispensed at least 1 study lens.
Measure: Number; unit: proportion
Units Other Than Participants: number of eyes
Arm/Group | Test (Senofilcon A) | Control (Etafilcon A)
Number analyzed (Participants) | 44 | 44
Number analyzed (number of eyes) | 88 | 88
proportion | 0.837 | 0.813

6. Primary Outcome: Binocular Contact Lens-Corrected Visual Performance Under Standard High Contrast Dim With Goggles
Description: as for outcome 1
Time Frame: 2-Week Follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Test (Senofilcon A) | Control (Etafilcon A)
Number analyzed (Participants) | 40 | 40
logMAR
  Standard High Contrast Dim with Goggles: Distance | 0.14 (0.109) | 0.13 (0.085)
  Standard High Contrast Dim with Goggles: Intermediate | 0.02 (0.095) | 0.00 (0.091)
  Standard High Contrast Dim with Goggles: Near | 0.18 (0.098) | 0.16 (0.101)

7. Primary Outcome: Binocular Contact Lens-Corrected Visual Performance Under Standard Low Contrast Bright
Description: as for outcome 1
Time Frame: 2-Week Follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Test (Senofilcon A) | Control (Etafilcon A)
Number analyzed (Participants) | 40 | 40
logMAR
  Standard Low Contrast Bright: Distance | 0.08 (0.093) | 0.07 (0.075)
  Standard Low Contrast Bright: Intermediate | 0.12 (0.075) | 0.10 (0.094)
  Standard Low Contrast Bright: Near | 0.25 (0.113) | 0.27 (0.119)

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study. Approximately 21-28 days per subject.
Description: All subjects dispensed at least 1 study lens.
Groups:
- Test: Subjects that wore the Test lens in either the first or second period of the study.
- Control: Subjects that wore the Control lens in either the first or second period of the study.
Arm/Group | Test | Control
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/44
Other Adverse Events (participants affected / at risk) | 0/44 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-25): https://cdn.clinicaltrials.gov/large-docs/24/NCT04189224/Prot_SAP_000.pdf